CLINICAL TRIAL: NCT06534333
Title: Can Ultrasonography Contribute to the Diagnosis of Patellofemoral Pain Syndrome?
Brief Title: Contribution of Ultrasonography in Patellofemoral Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, doctor, Ankara City Hospital Bilkent
Other Study IDs: Erololçok-dk-1
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life; Pain
Keywords: patellofemoral pain syndrome, ultrasonography, cartilage,
MeSH Terms: conditions — Pain; Patellofemoral Pain Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patellofemoral pain syndrome group
  Interventions: Other: Ultrasonography
- Group 2: Control group
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — musculoskeletal ultrasonography

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common cause of knee pain in adults younger than 60 years. . In this study, we aimed to evaluate the medial and lateral cartilage thickness the medial and lateral retinaculum thickness and the medial and lateral patellofemoral distance using ultrasonography and to compare with healthy controls. We also aimed to investigate the relationship between the measurements obtained in the PFPS group and pain intensity, functional scoring, and quality of life.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a common cause of knee pain in adults younger than 60 years. The prevalence of PFPS was found to be 7-28.2% and the incidence was 9.2%. In this study, we aimed to evaluate the medial and lateral cartilage thickness due to the possible relationship of PFPS with osteoarthritis, the medial and lateral retinaculum thickness as it is one of the static stabilizers of the patellofemoral joint, and the medial and lateral patellofemoral distance as it indicates patellar malposition, using ultrasonography and to compare with healthy controls. We also aimed to investigate the relationship between the measurements obtained in the PFPS group and pain intensity, functional scoring, and quality of life.This study is a non-randomized and non-blinded, cross-sectional clinical study with a control group. 54 eligible volunteers who applied to the physical medicine and rehabilitation outpatient clinic of Hitit University Faculty of Medicine.27 of the participants were patients diagnosed with unilateral PFPS, and 27 were healthy individuals without knee pain. Local ethics committee approved the study (2024/36) and informed consent was obtained from all participants.Participants were between the ages of 18-45. A positive result in at least one of the following four tests was considered diagnostic for PFPS, with pain occurring around or behind the patella and aggravated by at least one activity that placed load on the patellofemoral joint during weight bearing on the flexed knee. These tests 1) Medial or lateral patellar facet tenderness 2) Clark's test 3) Patellar apprehension test 4) Patellar tilt test. The inclusion criteria for the PFPS group were that the patients had knee pain for at least 3 month, unilateral pain, no history of knee surgery, no systemic disease, and no clinical symptoms of other knee pathologies other than PFPS. In order to exclude other pathologies that cause knee pain; patellar plica tests, Apley compression and distraction tests, McMurray tests, varus-valgus stress tests, anterior and posterior drawer tests, pivot shift and Lachman tests were performed. Those with positive results in these tests were excluded from the study.

The inclusion criteria for the control group were absence of anterior knee pain, no history of knee surgery, and no systemic disease.

Individuals with clinical symptoms related to other knee pathologies, history of trauma, history of patellar dislocation or subluxation, passive motion restriction in the knee joint, hip-spine related pain, the presence of any neurological disease affecting the extremities, inflammatory disease were excluded.

Detailed history and physical examination findings were recorded. The age, education level, marital status, height, weight, body mass index (kg/m2), duration of pain, dominant and affected extremity of all patients were recorded.

Pain levels at rest and during activity were measured using the Visual Analogue Scale (VAS).Kujala patellofemoral score was used to assess functional status of patients.Quality of life was evaluated with Short form-36 (SF-36). A B-mode ultrasound examination was performed by a radiologist with more than 5 years of experience using a Samsung RS85 Prestige (Medical Systems Corporation, Seoul, South Korea) with a high frequency (4-15 MHz) linear probe.The painful knee of the PFAS group and the non-dominant knee of the control group were evaluated by ultrasonography. The medial and lateral retinaculum thickness, medial femoro-patellar distance from the medial patellar edge to the medial femoral condyle, lateral patellofemoral distance from the lateral patellar edge to the lateral femoral condyle were measured in the axial plane with the patients in the supine position with the knee flexed 30°. The medial and lateral sides of the trochlear cartilage were measured in the axial plane with the knee in 140° flexion.

ELIGIBILITY:
Inclusion Criteria:

. The inclusion criteria for the PFPS group were that the patients had knee pain for at least 3 month, unilateral pain, no history of knee surgery, no systemic disease, and no clinical symptoms of other knee pathologies other than PFPS. In order to exclude other pathologies that cause knee pain; patellar plica tests, Apley compression and distraction tests, McMurray tests, varus-valgus stress tests, anterior and posterior drawer tests, pivot shift and Lachman tests were performed. Those with positive results in these tests were excluded from the study.

The inclusion criteria for the control group were absence of anterior knee pain, no history of knee surgery, and no systemic disease.

Exclusion Criteria:

Individuals with clinical symptoms related to other knee pathologies, history of trauma, history of patellar dislocation or subluxation, passive motion restriction in the knee joint, hip-spine related pain, the presence of any neurological disease affecting the extremities, inflammatory disease were excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1: Patients with patellofemoral pain syndrome Group 2: Healthy subjects without knee pain
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
trochlear cartilage thickness | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Çorum Erol Olçok Research and Training hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pacini P, Martino M, Giuliani L, Santilli G, Agostini F, Del Gaudio G, Bernetti A, Mangone M, Paoloni M, Toscano M, De Vito C, Ottonello C, Santilli V, Cantisani V. Patello-Femoral Pain Syndrome: Magnetic Resonance Imaging versus Ultrasound. Diagnostics (Basel). 2023 Apr 21;13(8):1496. doi: 10.3390/diagnostics13081496. PMID 37189597
- [Background] Crossley KM, Stefanik JJ, Selfe J, Collins NJ, Davis IS, Powers CM, McConnell J, Vicenzino B, Bazett-Jones DM, Esculier JF, Morrissey D, Callaghan MJ. 2016 Patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester. Part 1: Terminology, definitions, clinical examination, natural history, patellofemoral osteoarthritis and patient-reported outcome measures. Br J Sports Med. 2016 Jul;50(14):839-43. doi: 10.1136/bjsports-2016-096384. Epub 2016 Jun 24. No abstract available. PMID 27343241